CLINICAL TRIAL: NCT02095600
Title: Deep Brain Stimulation and Frameless Stereotactic Radiosurgery in the Treatment of Drug Resistant Invalidating Tremor
Brief Title: Radiosurgery for Drug Resistant Invalidating Tremor
Acronym: DB-SRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DB-SRS
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Severe Upper Limb Tremor Refractory to Medical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiosurgical thalamotomy (Experimental)
  Interventions: Radiation: Radiosurgical thalamotomy

INTERVENTIONS:
Radiation: Radiosurgical thalamotomy

SUMMARY:
Stereotactic lesioning of thalamus and basal ganglia for treatment of tremor is a well-known procedure which, prior to the introduction of deep brain stimulation, or DBS, was usually achieved using stereotactic surgical procedures.

Radiosurgery of invisible targets to treat movement disorders and intractable pain are still the domain of frame-based procedures, due to the need of a solid reference system registered to the anterior commissure-posterior commissure (AC-PC) line, which allows the use of stereotactic atlases.

In this study we want to utilize a mathematical method that uses atlas-derived stereotactic coordinates to perform frameless images-guided radiosurgery of such functional targets Particularly the aim of the present study is to investigate both the efficacy and the safety of the methodology to treat upper limb and hand tremor in elderly or in patients which are not ot susceptible of surgical procedures. For these reasons a dose escalation prospective trial have been designed.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by severe upper limb tremor refractory to medical therapy and who are candidate for a deep brain stimulation (DBS) procedure.
* Age: ≥ 18 years old
* Refusal of DBS procedure
* Written consent

Exclusion Criteria:

* Pregnancy
* Allergy to contrast medium
* DBS procedure susceptibility, if not refused

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Tremor control (improvement in FTMTRS and/or UPDRS motor) | 2 years
  Tremor control (improvement in Fahn Tolosa Marin Tremor Rating Scale, FTMTRS, and/or Unified Parkinson's Disease Rating Scale, UPDRS, motor)

SECONDARY OUTCOMES:
Targeting methodology validation (the lesions position, if present, will be compared to the treatment plan target position, deviations will be registered). | 2 years
The treatment safety will be evaluated. Toxicity will be registered according to NCI-CTCAE v3. | 2 years
  The treatment safety will be evaluated. Toxicity will be registered according to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 3,NCI-CTCAE v3.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Unit of Radiotherapy, Milan, Italy